CLINICAL TRIAL: NCT01568840
Title: Effectiveness of Global Postural Reeducation and Segmental Exercises on Function, Pain, and Quality of Life of Patients With Scapular Dyskinesis and Cervicalgia: A Randomized Clinical Study
Brief Title: Global Postural Reeducation and Segmental Exercises in Patients With Scapular Dyskinesis and Cervicalgia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Principal Investigator, Cinthia Santos Miotto de Amorim, Effectiveness of Global Postural Reeducation and Segmental Exercises on Function, Pain, and Quality of Life of Patients with Scapular Dyskinesis and Cervicalgia: A Randomized Clinical Study, Irmandade da Santa Casa de Misericordia de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 192/10
Record Dates: First submitted 2012-03-26; First posted 2012-04-02 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Scapular Dyskinesis; Cervicalgia
Keywords: Physical Therapy Modalities; Posture; Muscle Stretching Exercises; Dyskinesias; Neck pain
MeSH Terms: conditions — Neck Pain; Dyskinesias | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Global Postural Reeducation Group (Experimental): Global Postural Reeducation
  Interventions: Other: Global Postural Reeducation Group
- Segmental Exercises Group (Active Comparator): Segmental Exercises
  Interventions: Other: Segmental Exercises Group

INTERVENTIONS:
Other: Global Postural Reeducation Group — Sessions happened once a week for 10 weeks, lasting 60 minutes each and consisted in manual therapy maneuvers and global postural reeducation treatment.
  Other Names: Global Postural Reeducation; Stretching Exercises
  Arms: Global Postural Reeducation Group
Other: Segmental Exercises Group — Sessions happened once a week for 10 weeks, lasting 60 minutes each and consisted in segmental exercises (stretching and strengthening) treatment.
  Other Names: Segmental Exercises; Stretching and Strengthening Exercises
  Arms: Segmental Exercises Group

SUMMARY:
The purpose of this study is to assess the effectiveness of global postural reeducation relative to segmental exercises in the treatment of scapular dyskinesis with cervicalgia.

DETAILED DESCRIPTION:
Purpose: To assess the effectiveness of global postural reeducation relative to segmental exercises in the treatment of scapular dyskinesis with cervicalgia.

Methods: Participants with scapular dyskinesis and cervicalgia (n = 30) aged 18 to 65 years were randomly assigned to one of two groups: Global Postural Reeducation and Segmental Exercises(stretching and strengthening). Upper extremity was assessed using the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire. Function of the neck was estimated using the Neck Disability Index (NDI). Pain severity was measured using a Visual Analogical Scale. Health-related quality of life (HRQoL) was assessed using the Short Form (SF)-12. Assessments were conducted at baseline and after 10 weekly sessions (60 minutes each). Significance level was established at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Scapular Dyskinesis as per the SICK Scapula Rating Scale
* Chronic Cervicalgia (pain for at least three months)

Exclusion Criteria:

* Cervical Stenosis
* Myelopathy
* Prolapsed Inter-Vertebral Disk (as confirmed by magnetic resonance imaging),
* Winged Scapula due to lesions of the long thoracic nerve or spinal accessory nerve, (as documented by electromyography)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-02

PRIMARY OUTCOMES:
Function of the upper extremity | 10 weeks
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire was used to measure function of the upper extremity, where 0 corresponded to "no disability" and 100 corresponded to "most severe disability".

SECONDARY OUTCOMES:
Pain severity | 10 weeks
  The Visual Analogical Scale (VAS) was used to measure pain, where the left extremity corresponded to"no pain" and the right extremity, corresponded to"maximum pain".
Health-related quality of life (HRQoL) | 10 weeks
  The HRQoL was assessed using the Short Form (SF)-12, the abbreviated version of the SF-36, whose score ranges from 0 to 100, and higher scores reflect better quality of life.
Function of the neck | 10 weeks
  The Neck Disability Index (NDI) was used to measure fuction of the neck, whose score ranges from 0 to 50: disability (0-5); mild disability (5-14); moderate disability (15-24); severe disability (25-34) and totally disabled (35-50).

CONTACTS AND LOCATIONS:
Locations (1):
- Irmandade da Santa Casa de Misericordia de Sao Paulo, São Paulo, São Paulo, Brazil